CLINICAL TRIAL: NCT06337149
Title: Relationship Between Breathing and Attention in Children With Ondine Syndrome
Acronym: OndineCo
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230348; IDRCB: 2023-A00006-39 (Registry Identifier: IDRCB ANSM)
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Ondine Syndrome; Congenital Central Hypoventilation Syndrome (CCHS)
MeSH Terms: conditions — Sleep Apnea, Central; Congenital central hypoventilation syndrome | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: neuropsychological tests used usually in clinical practice (TEA-ch, NEPSY, BRIEF) and research (Conners 3, K-CPT II or CPT III, Flankers Task) — neuropsychological tests used usually in clinical practice (TEA-ch, NEPSY, BRIEF) and research (Conners 3, K-CPT II or CPT III, Flankers Task)

SUMMARY:
Congenital central hypoventilation syndrome (CCHS) is a rare disorder of autonomic and respiratory regulation that alters oxygen delivery to the brain. CCHS patients are at risk for broad neurocognitive deficits. Patients retain ventilatory activity when awake through a respiratory-related cortical network but the need to mobilise cortical resources to breathe lead to breathing-cognition interferences during cognitive tasks. The purpose of this study is to assess the relationship between breathing pattern and attention in CCHS children

DETAILED DESCRIPTION:
Congenital central hypoventilation syndrome (CCHS) is a rare genetic disorder caused by PHOX2B gene mutations. CCHS is characterized by hypoventilation and autonomic nervous system dysregulation and global dysautonomia necessitating artificial ventilation. CCHS increases the risk to develop neurocognitive deficiencies. Patients retain ventilatory activity when awake through a respiratory-related cortical network but the need to mobilise cortical resources to breathe lead to breathing-cognition interferences during cognitive tasks.

No study has focused on attentional abilities in CCHS pediatric population to highlight a specific attentional profile or to investigate the double task paradigm impact when attentional resources and management of spontaneous breathing are competing.

The aim of this study is to (i) Understand the link between spontaneous breathing and attentional functioning in CCHS children by comparing the evolution of breathing pattern relatively to the complexity of the attentionals tasks.

(ii) Characterize the attentional profil of CCHS patients by comparing attentional tasks performance of CCHS children versus control children (iii) Measure the impact of variables such as age and CO2 ventilatory response on attentional performances, by comparing attentional performances of the young patient group (< 50e p) to the attentional performances of older patient group (> 50e p) and studying the correlation between ventilatory response to CO2 and attentional performance (iv) Investigate the link between clinicals and behavioural tools regarding attentional and executive domains by studying the correlation between the cognitif test and inventories results Hypothese : attentional task could be link to a deficit in breathing function leading to hypoxemia and hypercapnia (alveolar hypoventilation).

Methode : compare CCHS patients performances and control group in neuropsychological tests used usually in clinical practice (TEA-ch, NEPSY, BRIEF) and research (Conners 3, K-CPT II or CPT III, Flankers Task).

Twenty children (age range : 6 to 16 years old) with CCHS and IQ > 70 and twenty control subjects in the same age range without neurodevelopmental disorder diagnosis will be enrolled.

Firstly, subjects of both groups will respond to a neuropsychological assessment including intellectual Wechsler scale (WISC V), instruction comprehension test (Nepsy II), a manual laterality test and attentional and executive assessment (TEA-ch + NEPSY II).

Secondarily, CCHS group assessment will be completed with a double task paradigm. Our protocol includes a simple task condition (the patient must remain still) and a double task condition (the patient respond to the flanker tasks and K-CPT II or CPT III).

Procedure : continuous recording of breathing parameters : oxygen saturation, exhaled PCO2 (PETCO2 with nasal cannula) and respiratory rate. Breathing respiratory parameters will be recorded during simple condition and double task condition. "

ELIGIBILITY:
Inclusion Criteria:

* children with CCHS (Ondine Syndrome) and IQ > 70, age from 6 to 16 years old, french speaking, informed consent signed by both parents and oral agreement in principle given by the subject.

Exclusion Criteria:

* IQ < 70

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Ondine Syndrome, children with CCHS
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Wechsler scale | 12 months
  Neuropsychological assessement
Nepsy II test | 12 months
  Neuropsychological assessement

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claude TABET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided